CLINICAL TRIAL: NCT05036473
Title: A Phase II Randomized, Parallel, Double-blind, Placebo-controlled, Multi-center Clinical Trial of the Efficacy and Safety of WD-1603 Carbidopa-Levodopa Extended-Release Tablets in Patients With Parkinson's Disease
Brief Title: A Study of the Efficacy and Safety of Carbidopa-Levodopa Extended-Release Tablets in Patients With Parkinson's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai WD Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WD-1603-2001
Record Dates: First submitted 2021-08-10; First posted 2021-09-05 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-08

CONDITIONS: Parkinson Disease
Keywords: WD-1603; Carbidopa-Levodopa Extended-Release Tablets
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: Active groups are the groups of Parkinson's disease patients who will receive WD-1603 tablets with 3 different dosages.
  Placebo group is the group of Parkinson's disease patients who will receive the placebo-matching tablets.
Who Masked: Participant, Investigator
Masking Description: The active drugs and placebo are labeled from the company and the study staff will give the drug to the subjects who are randomized.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 25/100mg treatment group (Experimental): 25/100mg WD-1603
  Interventions: Drug: WD-1603 Carbidopa-Levodopa Extended-Release Tablets
- 25/150mg treatment group (Experimental): 25/150mg WD-1603
  Interventions: Drug: WD-1603 Carbidopa-Levodopa Extended-Release Tablets
- 2x25/100mg treatment group (Experimental): 2x25/100mg WD-1603
  Interventions: Drug: WD-1603 Carbidopa-Levodopa Extended-Release Tablets
- placebo group (Placebo Comparator): placebo are tablets-matching with the same active groups.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: WD-1603 Carbidopa-Levodopa Extended-Release Tablets — Taking WD-1603 tablets or placebo orally three times a day, in the morning before meals, and the second and third medications will be taken after meals, once every 5 hours (±30 minutes).
  Other Names: WD-1603
  Arms: 25/100mg treatment group; 25/150mg treatment group; 2x25/100mg treatment group
Drug: Placebo — placebo tablets-matching the active groups.
  Other Names: Placebo of WD-1603
  Arms: placebo group

SUMMARY:
It is a phase II randomized, parallel, double-blind, placebo-controlled, multi-center clinical trial of the efficacy and safety of WD-1603 Carbidopa-Levodopa Extended-Release Tablets in patients with Parkinson's disease. The objective of the study is to access the safety and efficacy of WD-1603 carbidopa-levodopa extended-release tablets in patients with Parkinson's disease.

DETAILED DESCRIPTION:
Eligible subjects of the study will be randomly assigned into four groups at a ratio of 1:1:1:1: three treatment groups and one placebo group. The subjects will take trial drugs orally three times a day, in the morning before meals, and the second and third medications will be taken after meals, once every 5 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female patients with early Parkinson's disease who are over 30 years old and under 75 years old (including cut-off values).
2. Able to understand and willing to sign an informed consent form (ICF) voluntarily.
3. The diagnosis of Parkinson's disease complies with idiopathic Parkinson's disease (2015 version of MDS Parkinson's disease diagnostic criteria).
4. Modified Hoehn and Yahr Scale≥1, ≤2.5 points.
5. Agree to use medically acceptable contraceptive methods throughout the study and within 1 month after completing the study.

Exclusion Criteria:

1. Have a history of severe allergic reactions or allergies to levodopa or carbidopa.
2. Pregnancy or breastfeeding.
3. Diagnosed as atypical Parkinson's disease or any known secondary Parkinson's syndrome.
4. The investigator believes that the placebo treatment cannot be tolerated.
5. Acute psychosis or hallucinations, using any antipsychotic to treat psychosis or clinically obvious depression.
6. History of epilepsy or epilepsy.
7. The history of narrow-angle glaucoma.
8. Subjects with a history of malignant melanoma.
9. Patients with obvious cognitive impairment.
10. The investigator believes that there are clinically significant medical or surgical diseases and patients who are not suitable for participating in clinical trials.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2022-05-16 (Estimated); Study Completion 2022-09-16 (Estimated)

PRIMARY OUTCOMES:
To compare the changes from the baseline mean value before the study to the mean value on the 27th day of the study between each dose group and the placebo group. | 27 days- from the baseline to the 27th day
  To compare the changes from the baseline mean value before the study to the mean value on the 27th day of the study of the sum of MDS-Unified Parkinson's Disease Rating Scale-Part II (MDS-UPDRS-II) and MDS-Unified Parkinson's Disease Rating Scale-Part III (MDS-UPDRS-III) between each dose group and the placebo group. MDS-UPDRS-II is Motor Experiences of Daily Living, and MDS-UPDRS-III is Motor Examination. Each item is rated on a 5-point Likert-type scale (0-4), with higher scores suggesting more severe impairment.

SECONDARY OUTCOMES:
To compare the change from the baseline mean value before the study to the mean value on the 14th day of the study between each dose group and the placebo group. | 14 days-from the baseline to the 14th day
  To compare the changes from the baseline mean value before the study to the mean value on the 14th day of the study of the sum of MDS-Unified Parkinson's Disease Rating Scale-Part II (MDS-UPDRS-II) and MDS-Unified Parkinson's Disease Rating Scale-Part III (MDS-UPDRS-III) between each dose group and the placebo group. MDS-UPDRS-II is Motor Experiences of Daily Living, and MDS-UPDRS-III is Motor Examination. Each item is rated on a 5-point Likert-type scale (0-4), with higher scores suggesting more severe impairment.
To compare the change from the baseline mean value before the study to the mean value on the 14th and 27th days of the study between each dose group and the placebo group. | Day -21- -2, Day -1, Day 14, and Day 27
  Complete the MDS-Unified Parkinson's Disease Rating Scale-Part II (MDS-UPDRS-II) assessment on the morning of each visiting period.
To compare the change from the baseline mean value before the study to the mean value on the 14th and 27th days of the study of MDS-UPDRS-III between each dose group and the placebo group. | 14 days and 27 days-from the baseline to the 14th and 27th day
  During the screening period, an outpatient evaluation is performed before administration. In the other visit periods, 6 assessments of the MDS-Unified Parkinson's Disease Rating Scale-Part III (MDS-UPDRS-III) are carried out at the time point of the clinical trial administration.
To evaluate Cmax | 1 day- on the 28th day
  To evaluate Cmax (Maximum Plasma Concentration) of the pharmacokinetics of WD-1603 on the 28th day.
To evaluate Cmin | 1 day- on the 28th day
  To evaluate Cmin (Minimum Plasma Concentration) of the pharmacokinetics of WD-1603 on the 28th day.
To evaluate the AUC | 1 day- on the 28th day
  To evaluate the AUC (Area under the plasma concentration versus time curve) of the pharmacokinetics of WD-1603 on the 28th day.
To evaluate levodopa blood concentration fluctuation index. | 1 day- on the 28th day
  To evaluate levodopa blood concentration fluctuation index of WD-1603 on the 28th day.
  Plasma levodopa is summarized according to the blood sampling time point of the protocol; describe and compare the mean of the blood concentration of levodopa and carbidopa in each dose group, and calculate the fluctuation index ([Cmax-Cmin]/Cavg, Cavg= AUC0-t/t), where Cmax is Maximum Plasma Concentration, Cmin is Minimum Plasma Concentration, Cave is Average Plasma Concentration, AUC0-t is Area under the Plasma Concentration versus Time Curve Calculated from 0 to the Last Measurable Observation.
To evaluate reported adverse events (AEs) of WD-1603 in patients with Parkinson's disease. | 28 days-from baseline to the 28th day.
  AEs refer to all adverse medical events in clinical research subjects, which can be manifested as symptoms and signs, diseases, or abnormal laboratory tests, but they may not have a causal relationship with the study drug. The following must be recorded as AE when at least one of the following criteria is met: 1. Accompanying symptoms and signs; 2. The results of the examination require treatment measures (such as surgical intervention); 3. The result of the inspection leads to changes in the dosing schedule of the study drug (such as dose change, dosing delay, discontinuation) of the study. The following can be referred to do AE severity classification. 1 (Mild): Asymptomatic or mild; only clinically seen; 2(Moderate): Requires minor, or non-invasive treatment; 3 (Severe): Severe or medically significant but not immediately life-threatening; 4 (Life-threatening): Urgent treatment is needed; 5 (Death): Death related to adverse events.
To evaluate Beck Depression Inventory-II (BDI-II) scale of WD-1603 in patients with Parkinson's disease. | 28 days-from baseline to the 28th day.
  BDI-II scores are collected for safety assessment. BDI-II is a 21-item self-administered survey which is scored on a scale of 0-3 in a list of four statements arranged in increasing severity about a particular symptom of depression. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoxiong(Jim) Wei, MD,PhD, Study Director — Shanghai WD Pharmaceutical Co., Ltd.
Locations (1):
- Shanghai Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No